CLINICAL TRIAL: NCT06936189
Title: A Prospective, Multicenter, Single-Arm Objective Performance Criteria Clinical Trial Evaluating the Safety and Efficacy of a Single-Use Neurovascular Intravascular Shockwave Catheter and Intravascular Shockwave Therapy Device for Pretreatment of Calcified Lesions in the Extracranial Carotid Artery (CREATE Trial)） (Extended Follow-Up)
Brief Title: Prospective Trial of IVL for Calcified Carotid Lesions(CREATE Trial)(Extended Follow-Up)
Status: Recruiting | Type: Observational
Sponsor: Shanghai Bluesail Boyuan Medical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: LFBY-202502
Record Dates: First submitted 2025-04-12; First posted 2025-04-20 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Carotid Artery Stenosis
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Calcified Carotid Artery Stenosis Treated with IVL and Carotid Artery Stenting (CAS): All patients participating in this extended follow-up period are sourced from the registered clinical trial.

SUMMARY:
Purpose: To assess the long-term safety and efficacy of the intravascular lithotripsy system for pre-treatment of calcified carotid artery stenosis.

Design: Prospective, multicenter, single-arm study with an extended follow-up period.

Sample Size: 204 participants (based on the final number of cases enrolled in the registration trial).

Endpoints:

Primary: Surgical success rate (residual stenosis <30% after stenting). Secondary: Target lesion re-narrowing rate, target lesion revascularization rate, MAE rate, ipsilateral stroke rate, and MACCE rate at 3 and 6 months postoperatively.

Follow-Up: Participants will be followed up at 3 months ±15 days and 6 months ±30 days postoperatively.

Inclusion criteria:

All patients participating in this extended follow-up period are sourced from the registered clinical trial.

Ethics and Consent: The trial will be conducted in accordance with the Helsinki Declaration and Chinese regulations. Informed consent will be obtained from all participants or their legal guardians.

Sponsor: Shanghai Lanfan Boyuan Medical Technology Co., Ltd. Principal Investigator: Professor Huo Xiaochuan, Beijing Anzhen Hospital.

DETAILED DESCRIPTION:
### Detailed Description

This clinical trial evaluates the safety and long-term efficacy of a disposable neurovascular intravascular lithotripsy (IVL) catheter and intravascular lithotripsy treatment device for pre-treatment of calcified lesions in the extracranial segment of the carotid artery. The study is designed as a prospective, multicenter, single-arm trial （extended follow-up period）.

#### Study Population:

All patients participating in this extended follow-up period are sourced from the registered clinical trial.（The registered clinical trial:Participants aged 18-80 years with symptomatic (≥50%) or asymptomatic (≥70%) calcified carotid artery stenosis confirmed by CT angiography (CTA) and digital subtraction angiography (DSA) are eligible. Patients who have failed conventional balloon dilation and are planned for carotid artery stenting (CAS) will be included.）

#### Follow-Up: Participants will be followed up at 3 months ±15 days and 6 months ±30 days postoperatively. Assessments will include clinical evaluations, imaging studies (CT angiography or carotid ultrasound), and recording of adverse events.

* Endpoints:

  * **Primary Endpoint**: Surgical success rate defined as residual stenosis <30% after stenting.
  * **Secondary Endpoints**: Target lesion re-narrowing rate, target lesion revascularization rate, MAE (major adverse events) rate, ipsilateral stroke rate, and MACCE (major adverse cardiovascular and cerebrovascular events) rate at 3 and 6 months postoperatively.
* Ethical Considerations:

Informed consent will be obtained from all participants or their legal guardians. The study will be conducted in accordance with the Helsinki Declaration and local regulatory requirements.

ELIGIBILITY:
Inclusion criteria:

All patients participating in this extended follow-up period are sourced from the registered clinical trial.

Exclusion criteria:

none

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients participating in this extended follow-up period are sourced from the registered clinical trial.
Sampling Method: Non-Probability Sample
Enrollment: 204 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Target lesion re-narrowing rate | at 3 months and 6 months postoperatively
  Proportion of patients with ≥50% diameter stenosis at the target lesion, assessed by imaging at 3 and 6 months.

SECONDARY OUTCOMES:
Target lesion revascularization rate | at 3 months and 6 months postoperatively
  Incidence of repeat revascularization procedures at the treated lesion, evaluated at 3 and 6 months.
MAE (Major Adverse Events) rate | at 3 months and 6 months postoperatively
  Rate of major adverse events (death, myocardial infarction, stroke) within 3 and 6 months.
Ipsilateral stroke rate | at 3 months and 6 months postoperatively
  Incidence of stroke on the treated side, confirmed by clinical and imaging studies at 3 and 6 months.
MACCE (Major Adverse Cardio-Cerebrovascular Events) rate | at 3 months and 6 months postoperatively
  Composite rate of death, stroke, myocardial infarction, and revascularization at 3 and 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Beijing, China